**Official Title:** Randomized, Double-Blind, Vehicle-Controlled Pilot Study of the Efficacy and Safety of HylaCareTM in the Treatment of Acute Skin Changes in Patients Undergoing External Beam Radiotherapy for Tumors of the Breast.

NCT02165605

Protocol Date: May 07, 2014 – Version 5

STUDYTITLE: Randomized, Double-Blind, Vehicle-Controlled Pilot Study

oftheEfficacyandSafetyofHylaCare TMintheTreatment ofAcuteSkinChangesinPatientsUndergoingExternal

BeamRadiotherapyforTumorsoftheBreast.

PROTOCOLNUMBER: STU092012-058

PRINCIPALINVESTIGATOR: AsalShoushtariRahimiM.D.,M.S.

UniversityofTexasSouthwesternMedicalCenter

DepartmentofRadiationOncology

COInvestigators: AnnSpanglerMD

DepartmentofRadiationOncology

DanGarwoodMD

DepartmentofRadiationOncology

MarilynLeitchMD DepartmentofSurgery

RoshniRaoMD DepartmentofSurgery

BarbaraHaleyMD

DepartmentofMedicalOncology

ChulAhn,PhD Professor

DepartmentofClinicalSciences

5323HarryHinesBlvd Dallas,TX75390-9066 (214)648-9418

NUMBEROFPATIENTSTO

BETREATED: 30

ESTIMATEDSTARTDATE: 2013

TESTARTICLES: HylaCare TM (TestSerum)

Placebo(Control)

Vehicle

SPONSOR'SNAMEAND

ADDRESS: Hylaco,LLC

3401LeeParkwaySuite1504

Dallas,TX75219

.

| Version | Date |
|---------|---------------|
| 2 | March 6,2013 |
| 3 | August6,2013 |
| 4 | October3,2013 |
| 5 | May7,2014 |

This confidential information is provided to you as an investigat staff, and applicable institutional review board. It is understood without written authorization from Hylaco.

ororpotentialinvestigatortobereviewedbyyou,your thatthisinformationwillnotbedisclosedtoothers

### **TABLEOFCONTENTS**

### 1.INTRODUCTIONANDPURPOSE

### 2.BACKGROUND

2.1StudyObjectives

#### 3.STUDYDESIGN

### 4.STUDYPROCEDURES

- 4.1SubjectSelectionCriteria
- 4.2StudyDuration
- 4.3DataCollection
- 4.4ConcomitantMedication
- 4.5GeneralPlan
- 4.6TestArticleBlindingandAdministration

### **5.SOURCEOFRESEARCHMATERIAL**

- 5.1HylaCare <sup>™</sup>andVehicleControl
- 5.2ProperHandlingandStorage

### **6.EVALUATIONANDCONSENT**

- 6.1BaselineProcedures(Visit#BL)
- 6.2TableofBaselineandSubsequentAssessments
- 6.3FinalVisit
- 6.4InformedConsent

### 7.EFFICACYPARAMETERS

### 8.POTENTIALRISKS

- 8.1DefinitionofAdverseEvents
- 8.2SeverityofAdverseEvents
- 8.3StepstoDetermineifanAdverseEventRequiresExpeditedReporting

#### 9.DATAMONITORING

- 9.1StatisticalandAnalyticalMethods
- 9.2SubjectSafety
- 9.3MonitoringProcedures
- 9.4HandlingofDropoutsorPatientsLosttoFollow-Up
- 9.5DiscontinuationofPatientsfromStudy

### 10.PROCEDURESTOMAINTAINCONFIDENTIALITY

#### 11.PROTOCOLADMINISTRATION

- 12.1DiscontinuationofStudy
- 12.2ChangesinProtocol
- 12.3InstitutionalReviewBoard
- 12.4ReportingofData
- 12.5FinalReport,Publication,andProtectionofTradeSecrets

### 12.INVESTIGATORAGREEMENT

### 13.REFERENCES

### 1.INTRODUCTIONANDPURPOSE

Morethan 50% of all patients with cancer receives ome form of radiotherapy (RT), for curative or palliative purposes, during the course of their illness.

One of the dose-limiting effects of radiotherapy is the acute reaction that ionizing radiation induces in normal tissues. The severity of adverse events resulting from exposure to radiotherapy is, in general, related to age and general health as well as to treatment-related factors such as the area being treated, radiation dose per fraction, and the total dose administered.

Skintoxicityisthemostcommonacutesideeffectofradiotherapytothebreast,occurringinmore than 90% of patients. (1)

Thespecificpurposeofthistrialistodeterminewhetherthehyaluronancomponentsof HylaCare TM induceaneffectiveness response significantly greater than use of avehicle control which lacks those in gredients in the management of a cuteskin reactions to external beam radiotherapy.

### 2.BACKGROUND

Early-onsetadverseeventsoccurtotissuessoon aftertreatmentinitiationwithexternalbeam radiationtherapybegins. The emergence of such symptoms, when severe, can adversely affect the patient's quality of life, result intreatment interruptions, and can reduce patient compliance with the treatment regimen. Among the most common of these is skintoxicity, observed frequently in patients being treated for breast cancer. The onset of a cuteradio-epider mititis results in erythema, epilation, and epider molysis, with the skin in the treated are abecomingdry, pruritic, hypersensitive, easily irritated, and in the longer term, hyper-pigmented. With some forms of radiotherapy, treated skin may develop amo is treated for breast tumors may develop changes in skintexture. Most skin reactions resolve within a few weeks after treatment is completed, although the skin may remain slightly darker than pretreatment.

The present management of radiation-associated skin toxicity includes instructions for care of the affected areas and the use of skin care products which can combat symptoms, without inducing further skin ir ritation.

Attentionhasrecentlybeenfocusedontheeffe ctsofhyaluronan(HA)forthemanagementof radio-epithelitisandacuteskinreactions.Liguori etal.(2)reportedtheeffectsofhyaluronan serumwhenappliedtoskinsurfacesaffectedbyradiationtoheadandneck,breast,andpelvic tumors.Comparedtoamatchingplaceboserum,patientstreatedwiththeHAserumshoweda significantpostponementinthefirstsignsofacuteradio-epithelitisandareductioninthe severityofskinreactions.

ThepresentstudywillevaluatetheeffectivenessandsafetyofHylaCare Thinthemanagement ofacuteskinreactionstoextern albeamradiotherapy. HylaCare Theoretainsthepatented HylaSponge®System, composed of small and large molecular weight hyaluronan (hyaluronicacid) and polymerized HylaSponges of infinite molecular weight. Due to its structure and preparation, the HylaSponge Systemis designed to improve the controlled release and slow delivery of variousing redients. A Repeated Insult Patch Test (RIPT) with HylaCare Thin 30 volunteer subjects demonstrated no potential for eliciting either dermal irritation or sensitization (3).

Themajorproperties which make this biopolymer unique and valuable for skin care are:

- Itsabilitytobeloadedwith,andthenslowlyrelease,waterandavarietyofactive ingredients
- Extremelyhighwaterretention
- Thequalityofactingasa"secondskin", whichishydrated, protective, and biocompatible

HylaCare<sup>TM</sup>,formulatedasatopicalproduct,hassuper-hydratingproperties.Itcontainsskin moisturizerssuchaspurelowandhighmolecularweighthyaluronan,the HylaSponge<sup>®</sup>System,andsqualane.ThesecharacteristicsmakeHylaCare TM anexcellent candidateforuseintheskincareofpatientswhomaydevelopacuteskintoxicityassociated withtheuseofexternalbeamradiotherapy.

### 2.1StudyObjectives

Theobjectiveofthiscontrolledstudywillbe todeterminetheeffectivenessandsafetyof HylaCare<sup>TM</sup>inthemanagementofthesymptomsofacuteskintoxicityinducedbyexposureto externalbeamradiotherapyassociatedwiththetreatmentofbreastcancer.

Theprimarymeasuresofeffectivenesswillbe:

- 1. Physician'sFollow-UpEvaluation:assessingsignsandsymptomsateachirradiatedsiteat week5duringRTandat2weekspost-treatment:
- 2. Physician'sGlobalAssessment:assessingeachirradiatedsiteat5weeksofRTpriorto boostandat2weekspost-treatment

Asecondarymeasureofeffectivenesswillbe:

The patient's independent and separate assessment of the tolerance to radio the rapy of each treated site at Week 5 of radio the rapy and at 2 weeks after its completion.

AnadditionalmethodofevaluationwillbetheInvestigator's assessment (disease oriented team to do assessment) of the baseline and treatment timeline photos.

### 3.STUDYDESIGN

This will be a randomized, double blind, vehicl e-controlled evaluation of the effectiveness and safety of Hyla Care TM. The study will employ the patient as her own control, a commonly used methodfortheevaluation of topical dermatologic agents. Each patient will be randomized blindly as to whether the study serum will be applied to the medial or lateral portion of the treated breast, using the nipple as the dividing line (see Figure 1. below). The product and place bo will also be applied to the contra-lateral breast in the same fashion, as a further control. The study drug and place bo will be applied three (3) times daily, but not within 4 hours prior to radiation treatment. It is a well known fact that any cream or moisturizer that leaves a film on the breast prior toradiation treatment can cause a boluseffect which can increase surface dose to the breast worsening dermatitis. Thus, not opical agent should be applied to the breast 4 hours before radiation treatment.

Patientswillbeallocatedtothetreatmentusingarandomizedpermutedblock. Therewillbeno stratification. Patientswillberandomizedtoreceivetheinvestigational product to be applied to either the medial (inside) or lateral (outside) portion of the breast, a place boproduct will be used on the other side. Patients and clinical investigators will be blinded to the treatment assignments.

Patientswillalsocompletea dailylog,recordingdailyapplicationtimes.At,orpriorto,the firstradiotherapyvisit,thepatientwillbeprovidedwith3SetBagscontainingsufficient materialsfor3weeksoftreatment,orasneeded.PatientswillreceivemoreSetBagsat Week3andWeek5,orasneeded.Patientsan dinvestigatorswillnotknowwhichbottleof serumisstudyserumvs.placebo.Thebottleswillbelabeledwithanidentifyingcode showingthesubject'sinitialsplusapatientnumber,andanotherlabelindicatingwherethe serumistobeapplied(medialorlateralpartofthebreast).



Figure 1. Diagramshowing medial and lateral portions of breast sto be addressed. Application sthree (3) times per day will continue throughout the course of radio the rapy and for 24 weeks after its completion (end of study). On any treatment day, the rewill be an application of test and control products immediately after the radio the rapy. No application will be made within four (4) hours prior to radio the rapy.

HylaCare<sup>TM</sup>andamatching(inappearance,consistencyandodor)vehiclecontrolproductwill besuppliedinidenticallyappearingopaquebottles anddispensedaccordingtoarandomized codelistpreparedbytheStatistician.

Thispilotstudywillbeinitiallyconductedatonecenterwith 30 patients undergoing standard fractionation external beam radiotherapy.

Patientsenrolledinthisstudywillbethosewhoaretoundergocurativeorpalliative radiotherapyfortumorsofthebreast. Treatmentprescription willbe 50.4 Gyin 28 fractions with tangential beams, followed by a 10 Gyin 5 fr action electron or photon boost. Those who meet all selection criteria will have a history taken, undergoaphysical examination, and a baseline evaluation by the Investigator. This evaluation will describe the tumor location and symptoms, as well as the intended radiother apytreatment plan, dose, and duration of treatment. The radiation treatment protocol for each patient will be determined by the Radiation Oncologist.

After the commencement of radiotherapy, patients will be evaluated at Week 5, and at 2 weeks post-treatment, by one of the radiation on cology investigators who will examine and grade the breast for acutes kintoxicity changes using the NCIC-CTC version 4.0 scale. A second Investigator Grading Scale will also be used for evaluation. Evaluation of the changes will also include examination and questioning for ery thema, pruritis, pain, dryness, exfoliation, epilation, hyperesthesia, or other signs/symptoms at each site. A supra-clavicular field may be irradiated and may also be treated with Products A and B, but will not be assessed for dermatitis.

Atstudycompletion, both the Investigator and patient will, independently and separately, assess the overall dermatitis of their radiated breast and the contralateral (non-irradiated) breast.

1. GradingScale:NCIC-CTC

| Adverse Event | 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|---|
| Dermatitis radiation | Faint erythema or dry desquamation | Moderate to brisk erythema; desquamation patchy moist desquamation, mostly confined to skin folds and creases moderate edema | Moist desquamation in areas other than skin folds and creases bleeding induced by minor trauma or abrasion | Life-threatening<br>consequences; skin<br>necrosis or<br>ulceration of full<br>thickness dermis;<br>spontaneous<br>bleeding from<br>involved site; skin<br>graft indicated | Death |

### 2. InvestigatorGradingScale:

Gradethestatusofthemedialandlateralsidesoftheirradiatedskinas:

0=normalskin

1 = light epidermal irritation, consisting of the onset of erythema, possibly associated with slight edema

2=erythemawithdrydesquamation

3=wetdesquamation</=2cm

4=wetdesquamationfrom2.1-5cm

5=wetdesquamationfrom5.1-9cm

6=wetdesquamation>9.1cm

### **4.STUDYPROCEDURES**

### 4.1SubjectSelectionCriteria

PatientswillberecruitedbytheInvestigatorfromhis/heravailablepatientpopulation,orby referral.SelectedpatientsmustmeettheInclusionandExclusioncriteria:

### **InclusionCriteria**

- Female,age18orolder
- Diagnosisofbreastcancer
- Intactbreast(notsurgicallyabsent)
- Plannedfractionatedexternalbeamradiotherapytobedeliveredbyopposing, tangentialbeamsto50.4Gyin28fractionswithaplannedphotonorelectronboost of10Gyin5fractions(foratotalof33fractions)
- Abilitytounderstandandcomplywiththerequirementsofthisstudy
- AbilitytogiveInformedConsent
- Forsexuallyactivefemales,patientagreestouseacceptablemethodof birthcontrol

### **Exclusion Criteria**

- Womenwhoarepregnantorlactating
- Useofconcomitantskincarepreparationsatanyofthetreatedorcontrolportalareas tobeobserved
- Any infection or unhealed wound of the radiotherapy portal areas, or generalized dermatitis
- Severerenalfailure(serumcreatinine >3.0mg/dL)within6monthsofstudy registration

- Allergichistory,includinganaphylaxisorsevereallergiestoproductsinstudyserum orplacebo
- Plannedrelocationwhichwouldmakefollow-upvisitsimpossibleduringthecourseof thestudy
- CollagenvasculardiseasesuchasLupus,orscleroderma

### 4.2 Study Duration

Patientsselectedforthisstudywillbeundergoingradiotherapyforcurativeorpalliativetreatment withfractionatedexternalbeamradiotherapy tobedeliveredbyopposing,tangentialbeamsto 50.4Gyin28fractionswithaplannedphotonorelectronboostof10Gyin5fractions(totalof 33fractions). Patientswillbefollowedfor2weeksafterradiotherapyhasfinished, withafollow-upvisitsat2weekspost-treatment.

### 4.3DataCollection

Datawillbecollected(typewritten,orhandwrittenlegiblyinblackink)ontheappropriatecase reportformssuppliedbytheSponsor.

### 4.4 Concomitant Medications

Patients will be asked about changes in their medications (prescription, nonprescription, or herbals) during their participation including name of the drug, indication for use, dosage, date started and datestopped. Changes in medications will be recorded.

### 4.5GeneralPlan

The patient's overall treatment plan will be guided by her tumor type. In general, its planning steps will include:

- 1. Specialradiologicstudiesmaybeorderedtohelpplantheradiationtreatments
- 2. Devices(e.g.,breastboards,vaclok)maybefabricatedtomaintainproper positioningduringtreatment pertheradiationoncologist
- 3. Simulationx-rayswillbeperformedto ensureaccurateplanningofthesizeand directionoftheradiationtreatmentfieldsonaweeklybasis
- 4. Tattoosorothermarkerswillbeappliedtoensurethepropersetupfordailytreatment
- Custom-madeblocksmaybefabricated,basedonCTsimulation,toshieldnormal structures
- 6. Duringasetupsession,thefieldar rangementsandblockswillbecheckedforproper alignment
- 7. Ingeneral, the borders of the field are:
  - i. Superior:inferiortotheclavicle
  - ii. Lateral:mid-axillaryline
  - iii. Inferior:2cminferiortotheinfra-mammaryfold
  - iv. Medial:Mid-sternum

### 4.6TestArticleBlindingandAdministration

At,orpriorto,thefirstradiotherapyvisit,the patientwillbeprovidedwith3SetBagscontaining sufficientmaterialsfor3weeksoftreatment,orasneeded.PatientswillreceivemoreSetBags atWeek3andWeek5,orasneeded.EachSetBagwillcontaintwo(2)60mLbottlesof HylaCare<sup>TM</sup>,andtwo(2)i denticallyappearingbottlesofPlacebo(ControlVehicle).Both containerswillbelabeledwiththepatient'sinitials,studynumber,andlocationofskintobe covered(ie.rightlateralbreast,leftmedialbreast,etc.)Additionally,thepatientwillbe instructedastotheproperapplicationoftheserums,includingamount,location,coverage,

### andhandwashing. See "Patient Instructions", Form 8

The contents of each bottle (Hyla Care TM or Placebo) will have been determined by a computerized random assignments cheme, the code fo rwhich will be kept at the study site in a sealed envelope.

The radiotherapy nurse, research team or physician will instruct the patient as to the proper application method and ensure that the patient understands which container contents are to be applied to which site (see Figure 1 and Patient Instructions, Form 8). The patient will apply a sufficient amount of either Hyla Care or place ebo(asprescribedintheexperimentalrandomized design)to cover the entire marked surface of their irradiated skin area IMMEDIATELY ATTHE END OF THE TREATMENT SESSION. At this time the same treatment will be applied to the contralateral(non-irradiated)breast. The patient will make two other applications during the day ™andthe vehicle control. to ensure a total of three (3) daily applications of both Hyla Care No applications will be made within 4 hours before radiotherapy. The three (3) daily applications will continue throughout the course of radiotherapy and for 2 weeks after its completion. Adrawn dashed line on both treated and untreated breast, as seen in Figure 1 will determine areas for use of study serum and place bo.

### Thepatientwillalsobeinstructed:

- 1. Toapplyproductonlytotheareasidentifiedonbothbreasts immediatelyafterthe radiotherapysession,andthentwomoretimesthatday.
- 2. Onnon-treatmentdays,toapplytheproductthree(3)timesdaily
- 3. Nottouseotherskincareproductsonanyoftheradiotherapy-exposedskinareas
- 4. Toreportanygeneralizedreactionsoranylocalizedreactionsintreatmentareatothe investigatoratthenextdailysession,ormoreseverereactionsbytelephone(See Section8).
- 5. todiscontinueuseoftopicalagentsiftheydevelop>/=grade3dermatitis.

Suggestionsforpersonalcareoftheirradiatedtreatmentsitesmayinclude:

- 1. Avoidirritatingtheskin
- 2. Whenwashing,useonlylukewarmwaterandmildsoap,pattingthesurface dry
- 3. Avoidtheuseoftightclothing
- 4. Donotrub, scruborscratchtheskin
- 5. Avoidtheuseofheatingpadsoricepacks
- 6. Donotusepowders,creams,perfumes,deod orants,bodyoils,ointments,orlotions ontheirradiatedsurfaces
- 7. Avoiddirectsunexposure; if necessary, we arprotective clothing

### 5.SOURCEOFRESEARCHMATERIAL

### 5.1 HylaCare<sup>™</sup>(TestSerum)andPlace bo(VehicleControl)

HylaCare<sup>™</sup>(TestSerum)andPlacebo(VehicleControl)willbesuppliedinidenticallyappearing opaque60mLbottles.

HylaCare<sup>™</sup>containsthefollowingingredients: HylaSponge<sup>®</sup>System Water Xanthangum Hydroxyethylcellulose

### Squalane

EMTPolymer (Hydroxyethylacrylate,Sodiumacryloyldimethyl,Tauratecopolymer) Benzylalcohol-DHA(benzylalcohol,(dihydroaceticacid)

The Vehicle Control contains the above-noted in gredients except for Hyla Sponge System

### 5.2 ProperHandlingandStorage

- 1.Storetestarticlecontainersatroomtemperature
- 2.Donotfreeze

### **6.EVALUATIONSANDCONSENT**

Patients who meet all selection criteria will be enrolled in numerical sequence. The assigned number will correspond to the order in which they are enrolled. The following visits will occur:

| Visit# | Title | Time |
|--------|-----------------------|---------------------------------|
| BL* | BaselineEvaluation(s) | 0(Priortotreatment)orWeek1visit |
| 1 | Radiotherapy (RT) | Initiation |
| 2 | Follow-UpEvaluation | At5Weekspriortoboost |
| 3 | FinalEvaluation | 2weeksafterRTends |

### 6.1BaselineProcedures(Visit#BL)

AttheBaselineEvaluation,allenrolledpatientswillundergohistory,physical examination,andbaselinelaboratory/radi ologicalassessmentsdictatedbythe planoftreatmentforthetumortoundergoradiotherapy.

The Research Teamortreating Physician will complete these forms and actions:

- (Form1)InformedConsent(Form1)
- (Form2a/2b)Inclusion/ExclusionCriteria(Forms2A/2B)
- (Form3)PhysicianFollow-UpAssessmentForm3
- (Form4)DemographicsandHistoryForm4
- (Form5)GeneralPhysicalExaminationForm5
- (Form6)RadiotherapyTreatment
- (Form7)PatientDailyLog
- (Form8)PatientInstructions

### 6.2TableofBaselineandSubsequentAssessments

Assessment of all radiation-exposed skin areas will occur as directed in the table below following the initiation of radiotherapy and at 2 and 4 weeks after the completion of radiotherapy. These forms and activities will be completed or reviewed at each assessment:

<sup>\*</sup>BaselineEvaluationmayrequiremorethanonevisit.

| FORM/ACTION | Base<br>Line | Week<br>1 | Week<br>2 | Week<br>3 | Week<br>4 | Week<br>5<br>Priorto<br>boost | Week<br>6 | Week<br>7 | 2<br>weeks<br>post |
|---|---|---|---|---|---|---|---|---|---|
| InformedConsent | ٧ | | | | | | | | |
| Photography | ٧ | | | | | ٧ | | | ٧ |
| Inclusion/<br>ExclusionCriteria | ٧ | | | | | | | | |
| PhysicianFollow-<br>UpAssessment | | | | | | <b>V</b> ** | | | V |
| Demographics andHistory | ٧ | | | | | | | | |
| GeneralPhysical<br>Examination | ٧ | | | | | | | | |
| Concomitant<br>Medication | ٧ | review | review | review | review | review | review | review | review |
| Baseline<br>Assessment | ٧ | | | | | | | | |
| UrinePregnancy<br>Test | V*** | | | | | | | | |
| Radiotherapy<br>Treatment | | **** | | | | | | | |
| PatientDailyLog | | v | ٧ | Collect log page | v | Collect logpage | ٧ | v | V<br>collect<br>logpage |
| AdverseEvent | If<br>needed | If<br>needed | If<br>needed | If<br>needed | If<br>needed | If<br>needed | If<br>needed | If<br>needed | Ifneeded |
| PatientOverall<br>Evaluation | | | | | | V***** | | | ٧ |
| PhysicianGlobal<br>Assessment | | | | | | ٧ | | | ٧ |
| Patient<br>Completion | | | | | | | | | ٧ |

\*Photographsofpatient'sbreastspriortoradiationtherapy: Thebaselinephotoshouldbea close-upencompassingonlythebreasttobetreatedata45degreeobliqueanglewitharms elevatedoverthepatient'shead. Otherphotosshouldbeastraightfrontalviewofbothbreasts takenineitherastandingorseatedpositionwiththepatient'shandsonherhips, excludingher face. Boostareawillbelabeledpriortoweek5photoandaphotowillbetakenshowingtheboost area. Labeleachslideorphotographwiththedateandthepatientcasenumber. The labeled photographswillbestoredelectronically understudy specific patient folders.

#### 6.3 FinalVisit

This will occurat 2 weeks after the completion of radiotherapy. These forms and actions will be completed:

- Physician'sFollow-UpAssessmentForm3
   Describestheradiotherapytreatmentandprovidesatimelinetocompare irradiatedandnon-irradiatedbreastindications
- Physician'sGlobalAssessmentForm9

<sup>\*\*</sup>Separatephotowithboostdrawnonskin.

<sup>\*\*\*</sup>IfPatientisofchild-bear ingageandsexuallyactive

<sup>\*\*\*\*</sup>PriortofirstRadiationTherapy

<sup>\*\*\*\*\*</sup>Evaluationshouldbecompletedpriortoboo st,butPatientwillnotberemovedfromthe studyisthisiscompletedaftertheboost.

TobecompletedatWeek5priortoboostandalso2weekspostradiation

PatientOverallEvaluationForm10

Usedtoelicitpatientevaluationofprophylaxis

PatientCompletionForm11
 Finalcompilationofpatientdatauponstudycompletionordiscontinuation

### 6.4InformedConsent

Writtenconsentwillbeobtainedfromeachpatientpriortoenteringthistrialandwillbecome partofthepatient'spermanentstudyrecord. Eachpatientwillbeassuredthatstudy participationisvoluntaryandthatshemaywithdrawatanytime. Atthetimeofobtaining writtenconsent, the Investigator will advise patients of the experimental nature of Hyla Care the duration of the trial, alternate modes of prophylaxis, and prevalent adverse events that might occur and discuss willing ness to have photographstaken.

TM

### 7.EFFICACYPARAMETERS

Theprimarymeasuresofeffectivenesswillbe:

- Physician'sFollow-UpEvaluation(Form3):assessingsignsandsymptomsateach irradiatedsiteWeek5duringRTandat2weekspost-treatment
- Physician'sGlobalAssessment:assessingeachirradiatedsiteatWeek5RTpriortoboost andat2weekspost-treatment

Asecondarymeasureofeffectivenesswillbethepatient's independent and separate assessment of the tolerance to radiother apyofeach treated site at the completion of radiother apyand at 2 weeks after its completion.

AnadditionalmethodofevaluationwillbetheInvestigator's assessment (disease oriented team to do assessment) of the baseline and timeline photos.

Inaddition,otherlocal(irradiatedareas)symptoms/signs(e.g.,pain,tenderness,pruritus, dryness,epilation,hyperesthesia)andanygene ralizedadverseeventswillbeevaluatedonthe basisofNCICtoxicitycriteria <a href="http://ctep.cancer.gov/reporting/ctc.html">http://ctep.cancer.gov/reporting/ctc.html</a>.

Week5ofradiotherapyandatthe finalevaluation(2weekspost-treatment),theInvestigatorwill makeanoverallglobalassessmentofeffectivenessofradiationtoleranceofthetreatedbreast (medialandlateralbreastwillbescoredindividua lly). Thisassessmentwillbebaseduponthe Investigator's experience, comparing the skinappearance and symptomatology of the site with the normally expected degree of radiation damage for similar body sites. The overall result will be graded as:

0=poor (worsethantypical expectations)

1=fair(equalto.orslightlybetterthantypicalexpectations)

2=good (moderately better than typical expectations)

3=excellent(markedlybetterthantypicalexpectations)

The Investigator will also judge which of the paired sites (medial, lateral)) tolerated radiotherapy better, interms of: (1) symptoms experienced by the patient and (2) over all skin appearance. If investigator feels medial and lateral breast symptomatology equivalent, then this will be reported as such.

Independent of the Investigator, the patient will also assess which of the paired sites fared better in terms of: (1) symptoms experienced and (2) over all skin appearance, at the completion of radiother apy and 2 weeks post-treatment.

### 8. PotentialRisks

InvestigationalProduct:

Inprevious use of Hyla Careas a commercial product, no adverse events have been identified.

### PsychologicalStress:

Questionnaireswillbegiventothepatientasapartofthisstudy, which may make them feel uncomfortable. Patient can refuse to answer any of the questions, take a break or stop participating in this study at any time.

### LossofConfidentiality:

Anytimeinformationiscollected; there is a potential risk for loss of confidentiality. Every effort will be made to keep the patients information confidential; however, this cannot be guaranteed.

### Photographs:

Patientcouldfeelslightlyuncomfortableduringthephotographicsessionswhenaskedto positionthebodytotakethephotographofthebreastarea. Patients could be uncomfortable with standing still for an extended period of time or from turning their body invarious positions. They could be sensitive to the bright and repeating flashes from the camera, which can so me times cause head aches, irritation of the eyes, discomfort, after effects such as seeing spots, and in rare cases, could stimulate a migraine head acheore pileptics eizure.

Photographsincludeariskofidentification. Patientsprivacy will be protected to the greatest extent possible. Photos will be taken to exclude faces or any other identifying marks. Photos will only be identified by a unique subject identification number that contains no personal identifying information. For research purposes, photos may be used in scientific publications.

### RiskstoEmbryo,FetusorBreast-fedInfant:

Females:Forpatientswhoarepregnantorbreast-feedinganinfant,itispossiblethatthey mayexposetheunbornchildorinfanttorisks. Forthatreason,pregnantandbreast-feeding femalescannotparticipateinthestudy.Forpatientwhoareparticipatinginthisstudyand areofchildbearingageandsexuallyactive,resultsofaurinepregnancytestwillbe obtained,anditmustbenegativebeforeparticipatinginthestudy.Patienttakingpartinthis studyandwhoaresexuallyactive,mustusemedically-acceptablebirthcontrol (contraceptives)duringthestudy.Medically-acceptablebirthcontrol(contraceptives) includes:

- (1)Surgical sterilization (such as hysterectomyor "tubestied").
- (2)Approvedhormonalcontraceptives(suchasbirthcontrolpills,patchorring;Depo-Provera,Depo-Lupron,Implanon),
- (3) Barrier methods (such as condomordia phragm) used with a spermic ide (a substance that kills sperm), or
- (4)Anintrauterinedevice(IUD).

Patientwhobecomepregnantduringthisstudy, must notify the researchers immediately.

### **OtherRisks**

Theremaypossiblybeothersideeffectsthatareunknownatthistime.

Radiationexposuretoawoman's reproductive organs may harm an embryo orfetus. Also, if radioactive materials are used for certain types of scans, harm may come to an embryo, fetus, or an infant who is breast feeding.

Pregnancytestsperformedduringtheearlystagesofpregnancydonotalwaysreveal pregnancy. Therefore, radiation exposure that includes the reproductive organs will be limited to the first tendays after a woman who can be come pregnant has begun her most recent menstrual period. This is standard policy inclinics and hospitals within UT Southwestern. This policy applies unless there is an important medical reason requiring radiation outside this time frame.

RisksofRadiation-RadiationTherapy:

The radiation the rapy used in this research is the standard radiation the rapy, therefore, the risk of harminvolved is the same.

High-doseradiationtreatmentstoornearaman'stesticlesorawoman'sovariesmay produceharmfulchangesthatcouldbepassedontochildrenthroughaspermoranegg.

Women: Females able to have children should avoid be coming pregnant until after they have had three menstrual periods after the end of all radiation the rapy. After three menstrual periods, there is almost no risk of harmful changes to an egg.

Possiblesideeffectsofradiationtherapytothebreastinclude:

Likely(thesesideeffectsoccurin10%ormoreofpatients):

- Reddeningoftheskinduringtreatmentandforseveralweeksfollowing treatment
- Tanningoftheskinlastingmonthsandmaybepermanent
- Slightlysmallerbreastsizeorchangeinthewaythebreastlooks
- Tirednessandweaknessduringtreatmentandforseveralweeksfollowing treatment
- Swellingofthebreast
- Peelingoftheskinintheareatreatedwithradiation
- Mildpainatthesiteofradiationtreatmentrequiringoverthecounterpain Relievers.

LessLikely(thesesideeffectsoccurin3-9%ofpatients):

- Sorenessortightnessinmusclesofthechestwallunderthetreated breast
- Severepainatthesiteofradiationrequiringprescriptionpainrelievers

RarebutSerious(thesesideeffectsoccurinlessthan3%ofpatients):

- Cough
- Difficultybreathing
- Inflammationoftheheartmuscle
- Ribfracture
- Slightincreaseinriskforheartdiseaseforpatientswithcancerintheleftbreast
- Riskofdevelopinganothercancer

Ateachfollow-upassessment, patients will be evaluated for any adverse effects. These will be grouped as follows:

- 1.Localizedreactionsattheirradiatedsites
- 2.Otheradverseevents

 $The Investigator will enter details of any of these events on the Adverse Event Form. The {\tt the Investigator will enter details of any of these events on the Adverse Event Form.}$ 

duration, intensity, and any action taken will be recorded.

### 8.1DefinitionofAdverseEvent

Anadverseevent(AE)isanyuntowardmedicalo ccurrenceinapatientreceivingstudytreatment andwhichdoesnotnecessarilyhaveacausalrelationshipwiththistreatment.AnAEcan thereforebeanyunfavorableandunintendedsign(includinganabnormallaboratoryfinding), symptom,ordiseasetemporallyassociatedwiththeuseofanexperimentalintervention,whether ornotrelatedtotheintervention.

### 8.2SeverityofAdverseEvents

Allnon-hematologicadverseeventswillbegraded accordingtotheNCICommonTerminology CriteriaforAdverseEvents(CTCAE)version4.0.TheCTCAEv4isavailableat <a href="http://ctep.cancer.gov/reporting/ctc.html">http://ctep.cancer.gov/reporting/ctc.html</a>

IfnoCTCAEgradingisavailable, these verity of an AEisgraded as follows:

 $\underline{Mild(grade1):} the event causes discomfort without disruption of normal daily activities.$ 

Moderate(grade2):theeventcausesdiscomfortthataffectsnormaldailyactivities.

<u>Severe(grade3):theeventmakesthepatientunabletoperformnormaldailyactivitiesor significantlyaffectshis/herclinicalstatus.</u>

<u>Life-threatening(grade4):thepatientwasatriskofdeathatthetimeoftheevent.</u> Fatal(grade5):theeventcauseddeath.

### 8.3StepstoDeterminelfanAdverseEventRequiresExpeditedReporting

<u>Step11</u>dentify the type of adverse event using the NCI Common Terminology CriteriaforAdverseEvents(CTCAEv4).

Step2: GradetheadverseeventusingtheNCICTCAEv4.

<u>Step3:</u>Determinewhethertheadverseeventisrelatedtotheprotocoltherapy Attributioncategoriesareasfollows:

- Definite-TheAE is clearly related to the study treatment.
- Probable-TheAEis likely related tothestudytreatment.
- Possible–TheAE *may be related*tothestudytreatment.
- Unrelated—TheAE is clearly NOT related to the study treatment.

<u>Note</u>: This includes allevents that occur within 30 days of the last dose of treatment. Any event that occurs more than 30 days after the last dose of treatment and is attributed (possibly, probably, or definitely) to the agent(s) must also be reported accordingly.

Step4:Determinethepriorexperienceoftheadverseevent.

Expected events are those that have been previously identified as resulting from administration of the agent. An adverse event is considered unexpected, for expedited reporting purposes only, when either the type of event or these verity of the event is not listed in:

- thecurrentknownadverseevents listedintheAgentInformation Sectionofthisprotocol;
- thedrugpackageinsert;
- thecurrentInvestigator'sBrochure

The intensity of adverse events will be graded as mild, moderate, or severe to describe

these observations regardless of whether they are medical events, symptoms, or physical findings. For purposes of consistency, the following definitions of intensity are provided:

Mild: Easilytolerated, causes minimal discomfort and does not interfere

witheverydayactivities

**Moderate:** Causessufficient discomfort to interfere with normal

everydayactivities

**Severe:** Incapacitatingandpreventsnormaleverydayactivities

ASeriousAdverseEventis anyexperiencethatsuggestsasignificanthazard,contraindication, sideeffectorprecaution,andincludesanyexperiencewhich:

- isfatalorlife-threatening
- ispermanentlydisabling(i.e.,incapacitatingorinterferingwiththeabilitytoresume usuallifepatterns
- requiresin-patienthospitalizationorprolongationofhospitalization
- isasecondarycancer,oranoverdose

ForHylaCare TM, potentialadverseeventsmightincludeanallergicreaction. Althoughthis has not been observed in other clinical trials of hyaluronan-based agents, this product is hyaluronan derived from a biological source; hence, the Investigator should be aware of the possibility that the material theoretically could cause an allergic reaction.

AnySeriousAdverseEventFormshouldbefaxe d,thenemailedimmediatelytoHylaco (JanetL.DenlingerPhD,ChiefScientificOfficer2018861643/jdenlinger@hylaco.com)and JeanWu(214-645-8913/jean.wu@utsouthwestern.edu).Anydeathorseriousorunusual reactionistobereportedpromptly(within24hours)bytelephonetoDr.Denlinger(2018861562) or,inherabsence,toMorganHare(214559 6125),eventhoughitmaynotappeartoberelated toHylaCare TM.

Alladverseeventswillbereviewedatthemonthlyradiationoncologyresearchmeetingwhich includesradiationoncologistnotadheringtotheprotocol.

Anypreliminarytelephonereportofaserious adverseeventistobefollowedbyadetailed writtenreportsummarywithinthreeworkingdaysandmustincludecopiesofhospital/office recordsandotherdocumentswhenapplicable. Anadditionalfollow-upwrittenreportsummaryis tobeforwardedtoHylacowithin10daysofthe adverseevent. The Investigator will also notify his/herInstitutionalReviewBoard(IRB) of any deaths, serious or unexpected reactions.

Follow-upofalladverseeventswillbecontinu eduntiltheoverallclinicaloutcomehasbeen ascertained. Alldeaths, serious and non-serious adverseevents will be summarized in the report prepared for Hylacoafter the conclusion of the study.

<u>UTSWIRB:</u>SAEswillbecollectedfromthetimeconsentisgiven,throughoutthe treatmentperiod,anduntilsubject'sparticipationinthetrialhasendedorparticipants death.

Investigators and other site personnel must inform the UTSWIRB, of any serious or unexpected adverse events that occur in accordance with the reporting obligations of 21 CFR 312.32, and will concurrently forward all such reports to UTSW IRB. It is the responsibility of the investigator to compile all necessary information.

Ifanon-serious AE becomes serious, this and other relevant follow-up information must also be provided to UTSWIRB..

All SAEs have to be reported to UTSW IRB, whether or not considered causally related to the investigational product. All SAEs will be documented. The investigatoris responsible for informing the IRB and/or the Regulatory Authority of the SAE asperlocal requirements.

Non-serious adverse events will be collected from the time consent is given, throughout the treatment period and up to and including the 30 day follow-up period. After withdrawal from treatment, subjects must be followed-up for all existing and new AEs for 30 calendar days after the last dose of trial drug and/or until event resolution. All new AEs occurring during that period must be recorded (if SAEs they must be reported to the UTSW IRB). All study-related toxicities/ SAEs must be followed until resolution, unless in the Investigator's opinion, the condition is unlikely to resolved ue to the patient's underlying disease.

Allseriousadverseeventsmustbereportedtothe UTSouthwesternTELEPHONE LINE: (214) 633-1753 within 24 hours of the investigator's awareness of the occurrenceoftheevent. Allsafetyreportsshallbefaxedto(214)645-8913oremailtotheattentionoftheprojectmanager.

The following events meet the definition of UPR:

- Anyseriousevent(injuries,sideeffects,deathsorotherproblems), whichintheopinionofthePrincipalInvestigatorwasunanticipated, involvedrisktosubjectsorothers,andwaspossiblyrelatedtothe researchprocedures.
- 2. Anyserious accidentalor unintentional change to the IRB-approved protocol that alters the level of risk.
- 3. Any deviation from the protocol taken without prior IRB review to eliminate apparent immediate hazard to are search subject.
- 4. Anynewinformation(e.g.,publication,safetymonitoringreport, updatedsponsorsafetyreport),interimresultorotherfindingthat indicatesanunexpectedchangetotherisk/benefitratioforthe research.
- Anybreachinconfidentialitythatmayinvolverisktothesubjector others.

### 9.DATAMONITORING

### 9.1StatisticalandAnalyticalMethods

Thirtypatientswillberecruitedinthispilotst udy. Descriptive statistics will be computed to estimate the sample size needed for a future larger study if the study results looks promising.

Descriptive statistics will be obtained for baseline demographic, medical history,

physical examination, radiation the rapy treatment/dosimetry data.

Patientswillbeallocatedtothetreatmentusingarandomizedpermutedblock. Therewillbeno stratification.Patientswillberandomizedtoreceivetheinvestigationalproducttobeappliedto eitherthemedial(inside)orlateral(outside)portionofthebreast,aplaceboproductwillbeused ontheotherside. Patients and clinical investigators will be blinded to the treatment assignments. TheprimaryefficacyvariablesarethePhysici an'sFollow-UpEvaluation,tobeperformedat eachvisit, and the Physician's Global Assessment, to be performed at the end of radio the rapy and2(two)weeksafterthecompletionofradiotherapy.The key componentofthe Physician's Follow-UpEvaluationisthegrading, on an ordinal scale (0 to 5) NCIC-CTC, as well as the InvestigatorGradingScaleoftheirradiatedareaofthebreast.Thedatacollectedfromthe Physician'sFollow-UpEvaluationwillbegroupedintotwoparts, thosedatacollectedduring radiotherapyandthosedatacollectedfollowingthecompletionofradiotherapy. For each <sup>TM</sup>treatedsideandthecontrolsidewillbe patient,thedifferencebetweentheHylaCare determinedateachvisitduringradiotherapy. These differences will then be averaged for each patient. The significance of the mean difference among the patients will then be determined usingapairedt-testorWilcox onsigned-ranktest.Thedataobta inedduringtheperiodfollowing radiotherapywillbeanalyzedinthismanner.TheanalysisofthePhysician'sGlobal Assessmentwillalsobeperformedseparatelyatthecompletionofradiotherapyandattheend ofthefollow-upperiod. The comparison of the groups will be based on a paired t-testor Wilcoxonsigned-ranktest. Asecondary analysis will be performed to examine the possible influenceofbodyhabitus(BMI-breastsize)andradi ationhotspotsontheeffectivenessofthe HylaCare<sup>™</sup>prophylaxis.Allefficacyanalyseswillbebasedonamodifiedintent-to-treatpatient population. This population will be defined as allpatientswhocommenceradiotherapyandwho haveatleastoneon-treatmentvisit.

Thesecondaryefficacymeasureisthepatient's assessmentofthetolerancetoradiotherapy. Thesedatawillbecollectedattheendofradiotherapyandattheendofthefollow-upperiod.At eachtimepointthepatientwillbeaskedthreequestionsandwillrespondtoeachquestionby indicatingwhichproductwaspreferredorifthepatienthadnopreference.Foreachquestionthe analysiswillcompare,amongthosepatientswhohaveapreference,thepercentwhoprefer HylaCare TM tothepercentwhopreferthecontrol.Thecomparisonwillbebasedonanexact BinomialtestofthehypothesisthatthepercentwhopreferHylaCare TM is50%,thepercentthat correspondstothepatienthavingnopreferencebetweenHylaCare

Theevaluationofphotostakenduringthecourse ofradiotherapyrepresentsthethirdefficacy measure. These will be evaluated in a blinde dmanner by the disease oriented team (which may consist of breast surgeons, plastic surgeons, or medical on cologists) after the last patient complete spost-treatment week 2 follow-up and photo

Safetywillbeassessedthroughtherecordingofresponsesandotheradverseevents. All patients who under goprophylaxis will be included in the analyses. The adverse events will be classified using the NCIC-CTC version 4.0.

AllcomputationswillbeperformedusingStatisticalAnalysisSystem(SAS)software.

**Grading NCIC-CTC** 

| Adverse Event | 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|---|
| Dermatitis radiation | Faint erythema or | Moderate to brisk | Moist desquamation | Life-threatening | Death |
| | dry desquamation | erythema; | in areas other than | consequences; skin | |
| | | desquamation | skin folds and | necrosis or | |
| | | patchy moist | creases | ulceration of full | |
| | | desquamation, | bleeding induced by | thickness dermis; | |
| | | mostly confined to | minor trauma or | spontaneous | |
| | | skin folds and | abrasion | bleeding from | |
| | | creases moderate | | involved site; skin | |

| | | edema | | graft indicated | |
|---|---|---|---|---|---|
| Definition: A finding of | cutaneous inflammatory | reaction occurring as a r | esult of exposure to biolo | ogically effective levels of | f ionizing |

### InvestigatorGradingScale:

0=normalskin

1 = light epidermal irritation, consisting of the onset of erythema, possibly associated with slight edema

2=erythemawithdrydesquamation

3=wetdesquamation</=2cm

4=wetdesquamationfrom2.1--5cm

5=wetdesquamationfrom5.1-9cm

6=wetdesquamation>9.1cm

### 9.2SubjectSafety

Safety will be assessed through the recording of responses and other adverse events. All patients who undergo prophylaxis will be included in the analyses. The adverse events will be classified using the NC IC-CTC scale 4.0.

### 9.3MonitoringProcedures

The monitor will pay site visits to review each patient's Case Report Forms to help ensure completenessandaccuracyofdataentryspecified intheProtocol.AsrequiredbyGoodClinical Practices guidelines, clinical records will be reviewed to confirm that: (1) the case report forms are consistent with the Investigator's clinical records; (2) background clinical and laboratory data and concomitant medications are recorded on the account of test and control article use; and (4) there is timely, appropriate reporting of any adverse events.

Patientswillbeinstructedto discontinueuseoftopicalagentsiftheydevelop>/=grade3 dermatitis.

ThedataandsafetyMonitoringBoard/Committeeare:

- InternalDSMB/DSMC
- UTSWRadiationOnclolgyInvestigators
- ExternalDSMB/DSMC
- SimmonsCancerCenter

### 9.4HandlingofDropoutsorPatientsLosttoFollow-Up

All patients who meet the selection criteria will be considered evaluable for efficacy and safety. Every attempt will be made to ensure that all patients complete the required follow-up visits. Those not appearing will be telephoned and/or contacted by mail to ensure that they complete their visit schedule. The reason for all dropouts is to be specified by the Investigator on the PatientCompletionForm.

### 9.5 Discontinuation of Patients From Study

Participation in this study may be discontinued for any of the following reasons:

- adverseevents
- severeinter-currentillness

- administrativereasons
- patient'svoluntarydecisiontodiscontinueparticipation
- Investigator'sopinionthatitisnotinthepatient'sbestintereststocontinue

Any patient discontinued because of an adverse event will be followed for at least 4 weeks, or until the adverse event is resolved, or as otherwis e medically indicated. It is important that the reason and the date of discontinuation be reported on the Patient Completion Form. If at all possible, an assessment should be done at the time of with drawal.

Patients who failed to apply the test and control products as directed for more than 5 days during radiation will be removed from the study for noncompliance.

### 10. PROCEDURESTOMAINTAINCONFIDENTIALITY

Confidentialityofeachpatient'sidentitywillbemaintained. Asubjectnumberconsistingofthe patient'sinitialsandarandomnumberwillbeassignedtoeachpatientuponstudyentryandthat numberwillbeusedtoidentifythat patientforthedurationofthest udy. Onlythepatient'sinitials and numberswillbeused on case report forms as well as any study-related correspondence.

### 11.PROTOCOLADMINISTRATION

### 11.1DiscontinuationoftheStudy

Hylacoreserves the right to discontinue any study for administrative reasons at any time such as, but not limited to, a decision to discontinue further clinical investigation with the test article, improper conduct of the study by the Investigator, or inability to obtain the number of patients required by the Protocol. Reimbursements for reasonable expenses will be made if such action is necessary.

### 11.2ChangesintheProtocol

Any changes that may affect the scientific soundness of the investigation or the rights, safety, or welfare of the subjects must receive appropriate IRB approval prior to implementation. Any changes in this Protocol will require the express written consent of Hylaco.

#### 11.3InstitutionalReviewBoard

Prior to implementation of this study, the Protocol and Patient Consent Form must be reviewed and approved by a properly constitut ed Institutional Review Board (IRB). Noch angest hat relate to the safety or welfare of patients may be made to the consent form unless they are approved by the IRB and Hylaco. All major amendments to the Protocol and caser eport forms must also be approved by the IRB and by Hylaco.

### 11.4 ReportingofData

Allinformation required by the Protocolisto be provided, or an explanation given for omissions. All case report forms (CRFs) must be made available as soon as they are completed in order that the Study Monitor may verify the validity and completeness of those forms and permit transmittal of the data to the Sponsor.

AlldataandinformationontheseCRFsaretobeneatlyrecordedintypeorlegiblywrittenin blackinkforeaseofduplication,interpretationandanalysisbeforesubmissiontoHylaco.All correctionsontheCRFsshouldbecrossedoutneatlywithasingleline,andthenewentry initialedanddatedbythememberoftheInvestigator'sstaffmakingtilecorrection.Priorto forwardingtheCRFstoHylaco,theyshouldbereviewedforcompleteness,accuracy, and legibility by the Principal Investigator and the Study Monitor. He/shewillindicateby

signature on the appropriate forms that he/she has reviewed the data at each evaluation period.

### 12.0 REFERENCES

- (1) Reference: Topical Hyaluronic Acid vs. Standard of Care for the Prevention of Radiation Dermatitis After Adjuvant Radiotherapy for Breast Cancer: Single-Blind Randomized Phase III Clinical Trial. International Journal of Radiation Oncology\*Biology\*Physics Volume 83, Issue 4, 15 July 2012, Pages 1089–1094 Chelsea Pinnix, M.D., Ph.D.-, George H. Perkins, M.D., M.P.H.-, Eric A. Strom, M.D.-, Wendy Woodward, M.D., Ph.D.-,
- (2) Liguori, V., Guillemin, C., Pesce, G.F., Mirimanoff, R.O., and Bernier, J. (1997). Double-blind, randomized clinical study comparing hyaluronic acid cream to placebo in patients treated with radiotherapy. Radiotherapy and Oncology 42, 155-161.
- (3) Final Report: Repeated Insult Patch Test for HylaCare<sup>™</sup> Batch code lot # 34905R020711. Lab and 2-7-11.

APPENDIX A

**EVALUATIONS and ACTIONS** 

#### **BaselineVisit**

AttheBaselineEvaluation,allenrolledpatientswillundergohistory,physical examination,andbaselinelaboratory/radi ologicalassessmentsdictatedbythe planoftreatmentforthetumortoundergoradiotherapy.

The Research Teamortreating Physician will complete these forms and actions:

- (Form1)InformedConsent
- (Form2a/2b)Inclusion/ExclusionCriteria
- (Form3)PhysicianFollow-UpAssessment
- (Form4)DemographicsandHistory
- (Form5)GeneralPhysicalExamination
- ((Form6)RadiotherapyTreatment
- (Form7)PatientDailyLog
- (Form8)PatientInstructions

### 6.2TableofBaselineandSubsequentAssessments

Assessment of all radiation-exposed skin areas will occur as described in the table below following the initiation of radiotherapy and at 2 weeks after the completion of radiotherapy.

Theseformsandactivitieswillbecompletedorreviewedateachassessment:

| FORM/ACTION | Base<br>Line | Week<br>1 | Week<br>2 | Week<br>3 | Week<br>4 | Week<br>5<br>Prior<br>to<br>boost | Week<br>6 | Week<br>7 | 2<br>weeks<br>post |
|---|---|---|---|---|---|---|---|---|---|
| InformedConsent | ٧ | | | | | | | | |
| Photography | ٧ | | | | | ٧ | | | ٧ |
| Inclusion/<br>ExclusionCriteria<br>PhysicianFollow- | ٧ | | | | | | | | |
| UpAssessment | | | | | | V** | | | V |
| Demographics andHistory | ٧ | | | | | | | | |
| GeneralPhysical<br>Examination | V | | | | | | | | |
| Concomitant<br>Medication | v | review | review | review | review r | eview re | view re | view rev | iew |
| Baseline<br>Assessment | ٧ | | | | | | | | |
| UrinePregnancy<br>Test | <b>V</b> *** | | | | | | | | |
| Radiotherapy<br>Treatment | | **** | | | | | | | |
| PatientDailyLog | | ٧ | v | Collect log page | v | Collect log page | v | v | Collect log page |
| AdverseEvent | If<br>needed | If<br>needed | If<br>needed | If<br>needed | If<br>needed | If<br>needed | If<br>needed | If<br>needed | If<br>needed |
| PatientOverall<br>Evaluation | | | | | | <b>V</b> ***** | | | ٧ |
| PhysicianGlobal<br>Assessment | | | | | | ٧ | | | ٧ |
| Patient<br>Completion | | | | | | | | | ٧ |

Photographsofpatient'sbreastspriortoradiationtherapy:Thebaselinephotoshouldbea close-upencompassingonlythebreasttobetreatedata45degreeobliqueanglewitharms

elevatedoverthepatient'shead.Otherphotosshouldbeastraightfrontalviewofbothbreasts takenineitherastandingorseatedpositionwiththepatient'shandsonherhips, excludingher face.Boostareawillbelabeledpriortoweek5photoandaphotowillbetakenshowingthe boostarea. Labeleachslideorphotographwiththedateandthepatientcasenumber.The labeledphotographswillbestoredelectronicallyunderstudyspecificpatientfolders.

### **FinalVisit**

This will occurat 2 weeks after the completion of radiotherapy. These forms and actions will be completed:

- PhysicianFo Ilow-UpAssessmentForm3
   Describestheradiotherapytreatmentandprovidesatimelinetocompare irradiatedandnon-irradiatedbreastindications
- Physician'sGlobalAssessmentForm9
   TobecompletedatWeek5priortoboostandalso2weekspostradiation
  - PatientOverallEvaluationForm10
     Usedtoelicitpatientevaluationofprophylaxis
- PatientCompletionForm11
   Finalcompilationofpatientdatauponstudycompletionordiscontinuation

<sup>\*\*</sup>Separatephotowithboostdrawnonskin.

<sup>\*\*\*</sup>IfPatientisofchild-bear ingageandsexuallyactive

<sup>\*\*\*\*</sup>PriortofirstRadiationTherapy

<sup>\*\*\*\*\*</sup>Evaluationshouldbecompletedpriortoboo st,butPatientwillnotberemovedfromthe studyisthisiscompletedaftertheboost.

### **APPENDIXB**

### **FORMS**

### FORM 1

### CONSENT TO PARTICIPATE IN RESEARCH TEMPLATE

### Instructions

Please read this consent form carefully and take your time making a decision about whether to participate. As the researchers discuss this consent form with you, please ask him/her to explain any words or information that you do not clearly understand. The purpose of the study, risks, inconveniences, discomforts, and other important information about the study are listed below. If you decide to participate, you will be given a copy of this form to keep.

### Why is this study being done?

The study is being done to provide information about the effectiveness and safety of a product containing the patented HylaSponge<sup>®</sup>System and whether the use of this product reduces the tissue damage that results from radiotherapy treatment.

### Why is this considered research?

This is a research study because the HylaSponge<sup>®</sup> System is being compared to placebo when applied to the breast which is undergoing radiotherapy as part of treatment for cancer.

### The following definitions may help you understand this study:

- Double-blind means neither you nor the researchers will know which product you are receiving.
- Randomization means the products will be assigned by chance for application to either side of your breast.
- Standard medical care means the regular care you would receive from your personal doctor if you choose not to participate in this research.
- Researchers means the study doctor and research personnel at the University of Texas Southwestern Medical Center

### Why am I being asked to take part in this research study?

You are being asked to take part in this study because you are going to be receiving radiotherapy as part of your treatment for breast cancer.

### Do I have to take part in this research study?"

No. You have the right to choose whether you want to take part in this research study. If you decide to participate and later change your mind, you are free to stop participation at any time.

If you decide not to take part in this research study it will not change your legal rights or the quality of health care that you receive at this center.

### How many people will take part in this study?

We plan to have approximately 30 people participate in this study here at UT Southwestern.

### What is involved in the study?

If you volunteer to take part in this research study, you will be asked to sign this consent form and will have the following tests and procedures. Some of the procedures may be part of your standard medical care, but others are being done solely for the purpose of this study.

### **Screening Procedures**

To help decide if you qualify to be in this study, the researchers may ask you questions about your health, including medications you take and any surgical procedures you have had.

You may also have to fill out certain forms or have the following exams, tests or procedures:

### Visit 1:

- Demographic information (age, gender, race, ethnic origin, and skin type);
- Eligibility assessment and an explanation of study purposes and procedures;
- Complete medical history including vital signs (temperature, pulse, respirations, blood pressure), height, weight, physical exam, allergies;
- Record current medications, vitamins, or herbs that you are taking;
- Photographs of breast. At your first visit, and at Week 5, and 2 weeks post-radiation treatment, photographs will be taken. Photos will be taken to exclude faces or any other identifying marks. Photos will only be identified by a unique subject identification number that contains no personal identifying information. These photographs are part of the research. You will not be able to participate in the research if you do not want to have photographs taken.
- You will be randomized to receive the investigational product to be applied to either the medial (inside) or lateral (outside) portion of your breast, a placebo product will be used on the other side.
- You will be given a supply of the investigational product and placebo and instruction/demonstration for application.
- During participation, you will be asked to do the following:
- No application of any skin care product besides the study products
- No use of skin products that may affect the color of your skin, such as sunless tanning lotions;

### Study Medication/Intervention

You will be provided with the study products to apply three times a day to each side as designated according to your random assignment. Please be sure to wash your hands before and between each application of product/cream. The creams/products will be labeled with your Subject Number.

Products will be supplied by the sponsor. This part of the study will be blinded, that is, both products will be packaged identically by the sponsor and labeled product A and product B so that neither you, nor the investigator, nor the research team will be able to distinguish which Product is applied to areas of radiation exposure.

### Procedures and Evaluations during the Research

### **Study Visits**

- Every week during your radiation treatment you will be assessed by an Investigator.
- The Investigator will evaluate the status of your skin, comparing the medial (inside) to the lateral (outside), and determining an overall assessment of your skin's tolerance to the radiotherapy.
- At your first visit, and during Week 5, and 2weeks post-radiation treatment, photographs will be taken.
- On your last day of radiation, both you and your radiation oncologist will be asked to complete an assessment of your skin, giving you an opportunity to report how you felt the creams worked, and if the skin on one side of your breast fared better than the other side

### Study Visit 9: (2 weeks after last radiotherapy)

- The physician will examine your skin
- Photographs of your breast
- You will return of any unused investigational product, as well as empty containers

•

- We will ask you about your current medications and any changes in your medications
- We will ask you about any adverse events (side effects or medical problems) that you are having
- We will ask you to complete another patient assessment, giving you another opportunity to report how you felt the creams worked, and if the skin on one side of your breast fared better than the other side.
- Additionally, during the entire duration of this study, we will ask you to maintain a log describing when you applied the products/creams.

### • Restricted Therapies

- O Drugs, procedures, and/or treatments restricted during the course of this study include:
- Use of any skin products on the bilateral breast, unless directed by physician
- o Application of any additional skin care products besides the study products.

Please ask your doctor if you have any questions about the medications that you are taking.

The photographs, assessments, and measurements in this study are designed for research, not for medical purposes. They are not useful for finding problems or diseases. Even though the researchers are not looking at this information to find or treat a medical problem, you will be told if they notice something unusual. You and your regular doctor can decide together whether to follow up with more tests or treatment.

### How long can I expect to be in this study?

Your participation in this study will last about 11 weeks.

You can choose to stop participating for any reason at any time.

### What are the risks of the study?

### Study Procedure/Intervention

Because of your participation in this study, you are subject to the following risks: You should discuss these with the researchers and your regular health care provider.

### **Investigational Product**

In previous use of *HylaCare* TM, no adverse events have been identified.

### Psychological Stress

Some of the questions we will ask you as part of this study may make you feel uncomfortable. You may refuse to answer any of the questions, take a break or stop your participation in this study at any time.

### Loss of Confidentiality

Any time information is collected; there is a potential risk for loss of confidentiality. Every effort will be made to keep your information confidential; however, this cannot be guaranteed.

### **Photographs**

You could be slightly uncomfortable during the photographic sessions when asked to position your body to take the photograph of your breast area. You may be uncomfortable with standing still for an extended period of time or from turning your body in various positions. You may be sensitive to the bright and repeating flashes from the camera, which can sometimes cause headaches, irritation of the eyes, discomfort, after effects such as seeing spots, and in rare cases, could stimulate a migraine headache or epileptic seizure.

Photographs include a risk of identification. Your privacy will be protected to the greatest extent possible. Photos will be taken to exclude faces or any other identifying marks. Photos will only be identified by a unique subject identification number that contains no personal identifying information. For research purposes your photos may be used in scientific publications.

### Other Risks

There may possibly be other side effects that are unknown at this time. If you are concerned about other, unknown side effects, please discuss this with the researchers.

### How will risks be minimized or prevented?

You will be carefully screened prior to participation in this study to be sure that you do not have any conditions that would make it unsafe for you. You will be closely monitored during the study. You will be asked, at each visit, about how you are feeling and about any problems or changes in your health that you are having. If you have any adverse events (side effects) from the study products, your surgeon will discuss appropriate treatment with you.

### What will my responsibilities be during the study?

While you are part of this study, the researchers will follow you closely to determine whether there are problems that need medical care. It is your responsibility to do the following:

- Ask questions about anything you do not understand.
- Keep your appointments.
- Follow the researchers' instructions.
- Let the researchers know if your telephone number or address changes.
- Store study materials (containers of product) in a secure place at home away from anyone who is unable to read and understand labels, especially children.
- Tell the researchers before you take any new medication, even if it is prescribed by another doctor for a different medical problem or something purchased over the counter.
- Tell your regular doctor about your participation in this study.
- Report to the researchers any injury or illnesses while you are on study even if you do not think it is related.

## If I agree to take part in this research study, will I be told of any new risks that may be found during the course of the study?

Yes. You will be told if any new information becomes available during the study that could cause you to change your mind about continuing to participate or that is important to your health or safety.

### What should I do if I think I am having problems?

If you have unusual symptoms, pain, or any other problems while you are in the study, you should report them to the researchers right away. Telephone numbers where they can be reached are listed on the first page of this consent form.

If you have a sudden, serious problem, like difficulty breathing or severe pain, go to the nearest hospital emergency room, or call 911 (or the correct emergency telephone number in your area). Tell emergency personnel about any medications you are taking.

### What are the possible benefits of this study?

If you agree to take part in this study, there may or may not be direct benefits to you. The researchers cannot guarantee that you will benefit from participation in this research. You may benefit from a reduction in skin irritation, decreased inflammation, and improved healing, but this cannot be guaranteed.

We hope the information learned from this study will may provide a better understanding of the effects of HylaCare<sup>TM</sup> on irradiated skin.

### What options are available if I decide not to take part in this research study?

This is not a treatment study. You do not have to be part of it to get treatment for your elective procedure.

Will my insurance provider or I be charged for the costs of any part of this research study? No. Neither you, nor your insurance provider, will be charged for anything done only for this research study (i.e., the Screening Procedures, Experimental Procedures, or Monitoring/Follow-up Procedures described above).

However, the standard medical care for your condition (care you would have received whether or not you were in this study) is your responsibility (or the responsibility of your insurance provider or governmental program). You will be charged, in the standard manner, for any procedures performed for your standard medical care.

### What will happen if I am harmed as a result of taking part in this study?

It is important that you report any illness or injury to the research team listed at the top of this form immediately.

Compensation for an injury resulting from your participation in this research is not available from the University of Texas Southwestern Medical Center at Dallas.

You retain your legal rights during your participation in this research

### Can I stop taking part in this research study?

Yes. If you decide to participate and later change your mind, you are free to stop taking part in the research study at any time.

If you decide to stop taking part in this research study, it will not affect your relationship with the UT Southwestern staff or doctors. Whether you participate or not will have no effect on your legal rights or the quality of your health care.

If you are a medical student, fellow, faculty, or staff at the Medical Center, your status will not be affected in any way.

Your doctor may be a research investigator in this study. S/he is interested in both your medical care and the conduct of this research study. At any time, you may discuss your care with another doctor who is not part of this research study. You do not have to take part in any research study offered by your doctor.

## If I agree to take part in this research study, can I be removed from the study without my consent?

Yes. The researchers may decide to take you off this study if:

- Your medical problem becomes worse.
- The researchers believe that participation in the research is no longer safe for you.
- The researchers believe that other treatment may be more helpful.
- The sponsor stops the research for the safety of the participants.
- The sponsor cancels the research.
- You are unable to keep appointments or to follow the researchers' instructions.

### Will my information be kept confidential?

Information about you that is collected for this research study will remain confidential unless you give your permission to share it with others, or if we are required by law to release it. You should know that certain organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- Hylaco, LLC; <u>Disease Oriented Breast Team- Surgical Oncologist, Medical Oncologist, Plastic</u> surgeons
- Representatives of government agencies involved in keeping research safe for people; and
- The UT Southwestern Institutional Review Board.

Medical information collected during this study and the results of any test or procedure done may be included in your medical record and this information may be available to health care providers and authorized persons including your insurance company.

In addition to this consent form, you will be asked to sign an "Authorization for Use and Disclosure of Protected Health Information." This authorization will give more details about how your information will be used for this research study, and who may see and/or get copies of your information.

### Are there procedures I should follow after stopping participation in this research?

If you, the researchers, or the sponsor stops your participation in the research, you may be asked to do the following:

- Let the researchers know immediately that you wish to withdraw from the research.
- Return to the research center for tests that may be needed for your safety.
- Return any unused study materials, including empty containers.
- Discuss your future medical care, if any, with the researchers and/or your personal doctor.

### Whom do I call if I have questions or problems?

For questions about the study, Asal Rahimi MD 214 645-8525 For questions about your rights as a research participant, contact the UT Southwestern Institutional Review Board (IRB) Office at 214-648-3060.

### **SIGNATURES:**

### YOU WILL BE GIVEN A COPY OF THIS CONSENT FORM TO KEEP.

Your signature below certifies the following:

- You have read (or been read) the information provided above.
- You have received answers to all of your questions and have been told whom to call if you have any more questions.
- You have freely decided to participate in this research.
- You understand that you are not giving up any of your legal rights.
   You understand that a copy of this signed consent document, information about this study
   1 the results of any test or procedure done may be included in your medical record and this
   ormation may be available to health care providers and authorized persons including your
   urance company.

| Participant's Name (printed) | |
|--------------------------------------------|----------|
| Participant's Signature | Date |
| Name of person obtaining consent (printed) | |
| Signature of person obtaining consent | <br>Date |

### FORM 2A

| Test Article: HylaCare™ |
|-------------------------|
| Study No.: |
| Investigator's Name: |

### **INCLUSION CRITERIA**

| Patient No.: |
|---------------|
| Today's Date: |

| For the patient to be included in the study, all answers to the following questions 1-6 mus AND at least the answer to one part of question 7 must be checked YES | t be check | ked YES, |
|---|---|---|
| | YES | NO |
| 1. Is the patient 18 years or older? | | |
| 2. Is there a diagnosis of cancer of the breast? | | |
| 4. Will the planned radiotherapy be administered via tangential ports? | | |
| 5. Has the patient provided a prior written Informed Consent form t? | | |
| 6. Does the patient have the ability to understand ad comply with the requirements of this study? | | |
| 7. For sexually active females, one of the answers provided below must be "YES" | | |
| A. Has the patient agreed to use an acceptable method of birth control; or take oral contraceptives for at least one month prior to study and for the duration of the study? | | |
| b. Been sterile, infertile or otherwise incapable of becoming pregnant, or | | |
| c. been post-menopausal for at least one year? | | |
| Investigator's Signature: Date: | | |

### FORM 2B

| Test Article: HylaCare™ |
|-------------------------|
| Study No.: |
| Investigator's Name: |

### **EXCLUSION CRITERIA**

| Patient No.: |
|---------------|
| Today's Date: |

| For the patient to be included in the study, all answers to the following questions must be c | hecked N | 0 |
|---|---|---|
| | YES | NO |
| 1. Is the patient either pregnant or lactating? | | |
| 2. Is the patient using any medication that might interfere with the interpretation of the test article's effectiveness or safety? | | |
| 3. Will the patient be using any concomitant skin care preparations on any of the irradiated areas? | | |
| 4. Does the patient have any infection or unhealed wound in the intended radiotherapy skin port areas? | | |
| 5. Does the patient have any form of generalized dermatosis? | | |
| 6. Does the patient have any known disease to affect the skin healing process? (e.g. severe renal failure, etc.)? | | |
| 7. Does the patient have a history of anaphylaxis or multiple severe allergies? | | |
| 8. Does the patient have a history of allergy to avian-sourced protein products? (e.g., chicken, eggs)? | | |
| 9. Does the patient plan to relocate during the course of the study, making scheduled visits impossible? | | |
| 10. Does the patient have collagen vascular disease (Lupus, scleroderma)? | | |

Investigator's Signature: \_\_\_\_\_\_Date: \_\_\_\_\_

| Test Article: HylaCa | re™ | | F0F | om 2 | | |
|---|---|---|---|---|---|---|
| | | | FORM 3 | | Patient No.: | |
| Study No.: | | | | s Follow-Up<br>nent Form | | |
| Investigator's Name: | | | ] | | Today's Date: | |
| umberofweekso<br>weekspost-treatr<br>heck(X)signsors | ment<br>ympton | _<br>nsreporte | | theirradiatedsk | kina | reas: |
| Indication - | Right | breast | LeftBreast | | | Whichsideof |
| muication | Medi<br>al | Lateral | Medial | Lateral | | IRRADIATEDBREAST<br>ONLYisworse?<br>(M/L/equal) |
| Redness | | | | | | |
| Pain | | | | | | |
| Tenderness | | | | | | |
| Easilylrritated | | | | | | |
| Burning | | | | | | |
| Dryness | | | | | | |
| Hypersensitive | | | | | | |
| HairLoss | | | | | | |

Comments:

Other (describe)

[Form3,continued]

I. GradingNCIC-CTC

| Adverse Event | 1 | 2 | 3 | 4 | 5 |
|---|---|---|---|---|---|
| Dermatitis<br>radiation | Faint erythema or dry desquamation | Moderate to brisk erythema; desquamation patchy moist desquamation, mostly confined to skin folds and creases moderate edema | Moist desquamation in areas other than skin folds and creases bleeding induced by minor trauma or abrasion | Life-threatening<br>consequences;<br>skin necrosis or<br>ulceration of full<br>thickness dermis;<br>spontaneous<br>bleeding from<br>involved site; skin<br>graft indicated | Death |

Definition: A finding of cutaneous inflammatory reaction occurring as a result of exposure to biologically effective levels of ionizing radiation

### PleaseuseNCIC-CTCgradinganddiagrambelow:



II. Inaddition,usingtheInvestigatorGradingScal e,gradethestatusofthemedialandlateral sidesoftheirradiatedskinas:

0=normalskin

1 = light epider malirritation, consisting of the onset of erythema, possibly associated with slighted ema

2=erythemawithdrydesquamation

3= wetdesquamation</=2cm

4= wetdesquamationfrom2.1-5cm

**5=** wetdesquamationfrom5.1-9cm

6= wetdesquamation>9.1cm

| Investigator's Signature: | Date: |
|---------------------------|-------|

[Form3,continued]

| Medial: | squamation, note minimal a | nm maximal | amation size: |
|---|---|---|---|
| Lateral: ı | mm minimal x r | nm maximal | |
| Most severe desquam | nation is dry or wet | _? | |
| | ation visit: Describe any trea | - | |
| Other (describe): | | | |
| Please grade the curr<br>Right Breast | ent status of desquamation | healing at 2-week I | Post-Radiation visit: |
| Medial: | 1 = no evidence of | f healing (or worser | ning) |
| | 2 = Beginning of p | proliferation | |
| | 3 = Tissue granula | | |
| Lateral: | 4 = Re-epithelializ | ation | |
| Left Breast | | | |
| Medial: | 1 = no evidence of | f healing (or worser | nina) |
| | 2 = Beginning of p | | 9) |
| | 3 = Tissue granula | | |
| Lateral: | 4 = Re-epithelializ | | |
| - | ted any concomitant medicyes, please list below. | cation(s) since the | last visit, or has the medication |
| Medicatio | | Dose | indication |
| • | ted any adverse events sind<br>ow and complete Adverse E | | Yes: No: |
| I | | | |
| Investigator's Signatu | ıre: | | Date: |

| Test Article: HylaCare™ |
|-------------------------|
| Study No.: |
| Investigator's Name: |

# FORM 4 DEMOGRAPHICS AND MEDICAL HISTORY

| Patient No.: |
|---------------|
| Today's Date: |

| PATIENT DEMOGRAPHICS | | | |
|---|---|---|---|
| Date of Birth (mm/dd/yy): | <u></u> | SEX: | Female |
| Height (inches): | | Weight (poun | ds): |
| Race: | | | |
| Race: | | on: 5-Ot | por aposify |
| I-Wille, Z-Black, S-FI | spariic, 4–Asi | an, 5–Ou | ier, specify |
| BMI: Breast | Cup Size: | | |
| | _ | | |
| | MEDICAL I | | |
| System | (Check approp | Abnormal | If Abnormal, specify: |
| Allergies | 1101111011 | | ,,, |
| Drug Sensitivities | | | |
| Dermatologic | | | |
| HEENT | | | |
| Cardiovascular | | | |
| Pulmonary | | | |
| Gastrointestinal | | | |
| Renal | | | |
| Endocrine-metabolic | | | |
| GU Systems | | | |
| Musculoskeletal | | | |
| Peripheral Vascular | | | |
| Neurological | | | |
| Psychiatric | | | |
| Other | | | |
| Additional comments on Medical Histo | ory findings (if any | <b>/</b> ): | |
| Investigator's Signature: | | | Date: |

| Test Article: HylaCare™ Study No.: Investigator's Name: | FORM 5 GENERAL PHYSICAL EXAMINATION | | Patient No.: Today's Date: |
|---|---|---|---|
| PHYSICAL EXAMINATION | Normal | Abnormal | If Abnormal, specify: |
| Head and Neck | | | , <b>, , </b> |
| Skin and Mucosa | | | |
| Eyes | | | |
| Lymph Nodes | | | |
| Cardiovascular | | | |
| Chest and Lungs | | | |
| Abdomen | | | |
| Musculoskeletal | | | |
| Other | | | |
| Additional Comments (if any): | | | |

Date:\_\_\_\_\_

Investigator's Signature:

| Test Article: HylaCare™ Study No.: Investigator's Name: | FORM 6<br>RADIOTHERAPY<br>TREATMENT FORI | |
|---|---|---|
| Dateoffirstradiotherapysessi | on(mm/dd/yy):// | |
| MaximumHotspot: | | |
| Circlewhether6MV15MV18M | IVorMIXEDPHOTONSareused | |
| Ifmixedphotonsareused,plea | senoteweightingofeachphotone | energy. |
| #cc'sreceivinggreaterthan10 | 7%prescriptiondose: | |
| #cc'sreceivinggreaterthan110%prescriptiondose: | | |
| #ofcc'sofbreasttissueinthetangentialfield(breasttangentsincludingchestwallandribs) | | |
| Wholebreastradiationprescriptiondose:Maximumdose: | | |
| Whichbreastisbeingirradiated | d?RightLeft | |
| Wholebreastradiationprescri | ptiondose:Maxii | , |

Investigator'sSignature:

Date:

| Test Article: HylaCare™ |
|-------------------------|
| Study No.: |
| Investigator's Name: |

### FORM 7 **PATIENT DAILY LOG**

| Patient No.: |
|---------------|
| Today's Date: |

| Day (Date) | Morning (time of application) | Afternoon (time of application) | Evening (time of application) |
|---|---|---|---|
| Monday | · | | |
| Tuesday | | | |
| Wednesday | | | |
| Thursday | | | |
| Friday | | | |
| Saturday | | | |
| Sunday | | | |
| Day (Date) | Morning (time of application) | Afternoon (time of application) | Evening (time of application) |
| Monday | , | | |
| Tuesday | | | |
| Wednesday | | | |
| Thursday | | | |
| Friday | | | |
| Saturday | | | |
| Sunday | | | |
| Day (Date) | Morning (time of application) | Afternoon (time of application) | Evening (time of application) |
| Monday | The state of the s | | |
| Tuesday | | | |
| Wednesday | | | |
| Thursday | | | |
| Friday | | | |
| Saturday | | | |
| Sunday | | | |

Test Article: HylaCare™

Study No.:
Investigator's Name:

## FORM 8 PATIENT INSTRUCTIONS FORM

(to be given to the patient!)

| Patient No.: |
|---------------|
| Today's Date: |

You have been given two nearly identical pump containers of serum to be applied to your irradiated skin three times a day. The label on each container will tell you on which side to apply the serum, either medial (inside) or lateral (outside). The picture below shows you which container should be used on which location.

At Baseline visit or first week of treatment, at Week 3, Week 5 and 2 weeks post-treatment you will be given sufficient Set Bags as needed to complete the study.

Please outline the areas of skin that will be subject to irradiation. Note areas to be <u>included</u>instudywithaCIRCLE,andnoteareasoutsidestudyareawithanX.



Usediagramtoindicatewhichjartouseonwhichportionofbreast. Note:

- (1) The above-outlined areas, within the circles to indicate inclusion in the study, are the onestowhichthetestarticle products are beapplied.
- (2) The patient will be instructed how, where, and how much product to apply to each irradiatedskinarea.
- (3) The patient will also be instructed to apply these products only to the encircled areas, and not to apply any other skin care products to the sesites.



### **Application Methods**

Ensure that your hands are clean, then use the pump to dispense an adequate amount of serum. Apply enough serum to cover the entire area noted in the diagram. Wash your hands again, before switching to the other serum and applying to the other side. Do not use any other products on the treatment areas.

### Additional Information

Apply serums three times a day, every day, but **ensure that you don't apply anything to your skin within 4 hours before your radiotherapy appointment.** 

Ensure that you apply the serums IMMEDIATELY AFTER radiotherapy treatment. Apply only to the area identified for prophylaxis.

Report any reactions (general or localized) to the investigator at the next daily session, or more severe reactions by telephone.

Suggestions for personal care of the irradiated skin

- 1. Avoid irritating the skin
- 2. When washing, use only lukewarm water and mild soap, patting the surface dry
- 3. Avoid the use of tight clothing
- 4. Do not rub, scrub or scratch the skin
- 5. Avoid the use of heating pads or ice packs
- 6. Do not use powders, creams , perfumes, deodorants, body oils, ointments or lotions on the irradiated surfaces
- 7. Avoid direct sun exposure, if necessary, wear protective clothing

| Study No.: |
|----------------------|
| Investigator's Name: |

# Form 9 PHYSICIAN'S GLOBAL ASSESSMENT FORM

| Patient No.: |
|---------------|
| Today's Date: |

**Note:** ThisformshouldbecompletedatWeek5 priortoboostandattheendofstudy (2weeksaftercompletionofRT).

Pleasemakeanoverallglobal assessmentoftheeffect ivenessofradiationskin toleranceofbothsidesof theirradiatedbreasttissue.Basedonyourjudgmentand pastexperience,comparetheskinappearanceandpatient'sreportedsymptomatology foreachsideofthebreast,andforeachbreas t(testsubstance-treatedandvehicle control-treated)withthenormallyexpected degreeofradiationdamageforsimilarbody sites.Gradeyouroverallimpressionas:

0=poor(worsethantypicalexpectations)

1=fair(equalto,orslightly betterthantypicalexpectations)

2=good(moderatelybetterthantypicalexpectations)

3=excellent(markedlybette rthantypicalexpectations)

Pleasecomparethetwoirradiat edsites.Inyouropinion, whichskinsitefaredbetter, basedonsymptomsexperienc ebythepatientandoverallskinappearance?

| Medial:l<br>LeftBreast | Lat | eral: | _EqualTole | rance: |
|---------------------------|-------|-------|----------------|------------|
| | Later | al: | _Equal | Tolerance: |
| Comments: | 1 | ) ! | ( <sub>\</sub> | |
| | Right | | Lef | ft |
| Investigator's Signature: | | | | Date: |

RightBreast:

| Test Article: HylaCare™ |
|-------------------------|
| Study No.: |
| Investigator's Name: |

# FORM 10 PATIENT'S OVERALL EVALUATION FORM

| Patient No.: |
|---------------|
| Today's Date: |

Date:

**Note:** The patient should complete this question na ire at Week 5 prior to boost and at the final visit (2 weeks a fter the completion of RT).

### InstructionstothePatient

Youhavenowcompletedyour prescribed course of radiot herapy administrated to your breast

| Please compare the two sides (medial [inner] and lateral [out er]) of your irradiated breastwhichwereexposedtoradiation. |
|---|
| In terms of any localized skin reactions you have experiences throughout your radiotherapy(suchasredness,so reness,itching,orothers),whichsideoftheirradiated breastdoyoubelievefaredbetter. Medialbetterthanlate ral(innerbetterthanouter)Nodifferencebetweenmedial(inner)andlateral(outer) |
| Whichsideoftheirradiatedbreasthasmain tainedanoverallappearanceclosesttoits appearancebeforera diotherapybegan? Medial(inner) Lateral(outer) Nodifferencebetweenmedial(inner)andlateral(outer) |
| Doyouhaveanypreferencesbetween theserumsappliedtoyourskin? Prefertheproductapplie dtomedialside(inner) Prefertheproductapplie dtolateralside(outer) Nopreferencebet weenthetwoproducts |
| Right |
| Ifyoudidpreferoneproductover theother,pleaseexplainwhy: |

Investigator's Signature:

| Test Article: HylaCare™ |
|-------------------------|
| Study No.: |
| Investigator's Name: |

### FORM 11 **PATIENT COMPLETION FORM**

| Patient No.: |
|---------------|
| Today's Date: |

| Note: To be completed at the final visit, or upon discontinuation from | the study. | |
|---|---|---|
| Subject Overview Did the patient experience any side effects from the study agent? | Yes: | No: |
| If yes, complete Adverse Event Form | | |
| 2.Study Completion Did the patient complete the entire study? | Yes: | No: |
| If no, complete information below. | | |
| 3.Discontinuation from Study Date of withdrawal (mm/dd/yy):/ | | |
| Reason for withdrawal (check and explain)Adverse Event:Did not meet protocol criteria:Unreliable:Lost to follow-up/moved: Subject requested discontinuation: Other: | | |
| Explain (in detail, as needed) | | |
| I have reviewed and evaluated the information provided in these cas represents the patient's clinical progress in the study. | | |
| Investigator's Signature: | Date: | |